CLINICAL TRIAL: NCT02028065
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Incidence of Hypersensitivity After Repeated Single Dose Administration of Sugammadex (MK-8616) in Healthy Subjects
Brief Title: A Study to Evaluate the Incidence of Hypersensitivity After Administration of Sugammadex in Healthy Participants (MK-8616-101)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8616-101; 2013-004640-37 (EudraCT Number)
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Hypersensitivity; Anaphylaxis
Keywords: reversal of neuromuscular blockade
MeSH Terms: conditions — Hypersensitivity; Anaphylaxis | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugammadex 4 mg/kg (Experimental): Administration of 3 single IV doses of sugammadex 4 mg/kg, with an approximately 5-week washout between Dose 1 and Dose 2 and between Dose 2 and Dose 3
  Interventions: Drug: Sugammadex
- Sugammadex 16 mg/kg (Experimental): Administration of 3 single IV doses of sugammadex 16 mg/kg, with an approximately 5-week washout between Dose 1 and Dose 2 and between Dose 2 and Dose 3
  Interventions: Drug: Sugammadex
- Placebo (Placebo Comparator): Administration of 3 single IV doses of placebo, with an approximately 5-week washout between Dose 1 and Dose 2 and between Dose 2 and Dose 3
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sugammadex — Sugammadex 4 mg/kg or 16 mg/kg administered as a single IV bolus over 10 seconds
  Arms: Sugammadex 16 mg/kg; Sugammadex 4 mg/kg
Drug: Placebo — Placebo administered as a single IV bolus over 10 seconds
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the potential for hypersensitivity symptoms upon repeat exposure to sugammadex. Healthy participants will be randomized to one of three treatment arms: sugammadex 4 mg/kg, sugammadex 16 mg/kg or placebo. Participants will receive 3 single intravenous (IV) doses of their randomized treatment, with an approximately 5-week washout between Dose 1 and Dose 2 and between Dose 2 and Dose 3. Participants will be confined at the study center from the day before each dose until completion of the 24-hour post dose assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-breast feeding female
* Females of childbearing potential must have a serum β-human chorionic gonadotropin (β-hCG) level consistent with non-pregnant state and agree to use (and/or have their partner use) two acceptable methods of birth control beginning at screening, throughout the trial (including washout intervals between treatment periods) and until after the post-study follow-up visit
* Females not of childbearing potential must be either a) postmenopausal (have not had a menstrual period for at least 1 year and have a follicle stimulating hormone [FSH] value in the postmenopausal range) or b) surgically sterile (i.e., have had hysterectomy, oophorectomy or tubal ligation)
* In good health based on medical history, laboratory tests and other assessments
* Body Mass Index (BMI) ≥19 and ≤32 kg/m^2
* Non-smoker or smokes ≤10 cigarettes/day or equivalent (2 pipes/day, 1 cigar/day) and agrees not to smoke while confined at the study center

Exclusion Criteria:

* Mentally or legally incapacitated, has significant emotional problems at the time of screening visit or expected during the conduct of the trial or has a history of clinically significant psychiatric disorder of the last 5 years
* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological abnormalities or diseases
* History of cancer (malignancy)
* History of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* Has had major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to screening
* Has participated in another investigational trial within 4 weeks prior to screening
* Is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of the initial dose of trial drug, throughout the trial (including washout intervals between treatment periods), until the post-study follow-up visit
* Has received subcutaneous or sublingual immunotherapy within the past 1 year
* Consumes >3 glasses of alcoholic beverages per day
* Consumes excessive amounts, defined as >6 servings of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 12 months
* Has a recollection of previously receiving sugammadex, Bridion™, SCH 900616, ORG 25969, or MK-8616
* History of chronic urticaria or angioedema
* Is or has an immediate family member (spouse or children) who is a member of investigational site or sponsor staff directly involved with this trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 382 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2014-07-01 (Actual); Study Completion 2014-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Min KC, Bondiskey P, Schulz V, Woo T, Assaid C, Yu W, Reynders T, Declercq R, McCrea J, Dennie J, Adkinson F, Shepherd G, Gutstein DE. Hypersensitivity incidence after sugammadex administration in healthy subjects: a randomised controlled trial. Br J Anaesth. 2018 Oct;121(4):749-757. doi: 10.1016/j.bja.2018.05.056. Epub 2018 Aug 23. PMID 30236237
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=8616-101&kw=8616-101&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant who was randomized to sugammadex 16 mg/kg instead received 3 doses of placebo and completed study. This participant appears in sugammadex 16 mg/kg column in Participant Flow period "Randomization through Start Treatment" and in placebo column in period "Treatment through Study Completion."
Groups:
- Placebo: Administration of 3 single intravenous (IV) doses of placebo, with an approximately 5-week washout between Dose 1 and Dose 2 and between Dose 2 and Dose 3
Period: Randomization Through Start Treatment
Arm/Group | Placebo | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg
Started | 76 (Randomized) | 154 (Randomized) | 152 (Randomized)
Completed | 75 | 151 | 149
Not Completed | 1 | 3 | 3
Not completed — Not treated | 1 | 3 | 3
Period: Treatment Through Study Completion
Arm/Group | Placebo | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg
Started | 76 (Includes 1 participant randomized to sugammadex 16 mg/kg who actually received placebo) | 151 | 148 (Does not include the 1 participant randomized to sugammadex 16 mg/kg who actually received placebo)
Received First Dose | 76 | 151 | 148
Received Second Dose | 69 | 140 | 138
Received Third Dose | 64 | 136 | 134
Completed | 64 | 136 | 134
Not Completed | 12 | 15 | 14
Not completed — Lost to Follow-up | 2 | 4 | 6
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 4 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 3
Not completed — Adverse Event | 3 | 3 | 5

BASELINE CHARACTERISTICS:
Population: All participants as treated (APaT) - All randomized participants who received at least one dose of study treatment, with each participant included in arm corresponding to treatment actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Total
Number analyzed (Participants) | 76 | 151 | 148 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (10) | 39 (11) | 38 (11) | 38 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 83 | 80 | 198
  Male | 41 | 68 | 68 | 177

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adjudicated Symptoms of Hypersensitivity
Description: The investigator or designated clinician performed a targeted hypersensitivity assessment (THA) in each participant at 0.5, 4 and 24 hours after each dose for each dosing period. The THA could also be performed at other times if possible hypersensitivity signs were observed. The THA included elicitation of symptoms as well as examination of the participant, covering neurologic, pulmonary, cardiovascular, gastrointestinal and dermatologic domains. Each potential hypersensitivity case identified by the presence of any sign or symptom in a pre-defined list of hypersensitivity signs and symptoms that were found through the THA was reviewed by an independent, blinded adjudication committee, which determined whether the referred case was a case of hypersensitivity (yes/no). In addition, all adverse events (AEs) occurring in study were reviewed for terms associated with hypersensitivity or anaphylaxis, and could also result in referral to the adjudication committee for evaluation.
Time Frame: Up to approximately 28 days after last dose (approximately 14 weeks)
Population: APaT - All randomized participants who received at least one dose of study treatment, with each participant included in arm corresponding to treatment actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg
Number analyzed (Participants) | 76 | 151 | 148
percentage of participants | 1.3 [0.0 to 7.1] | 6.6 [3.2 to 11.8] | 9.5 [5.3 to 15.4]
Statistical Analysis 1: Comparison: Placebo vs Sugammadex 4 mg/kg; Planned sample size of 150 participants in each sugammadex group (4 mg/kg and 16 mg/kg) allowed estimation of adjudicated hypersensitivity in each sugammadex group with a 95% confidence interval with a half-width between 1.2 and 4.2 percentage points. Calculation, based on method of Clopper and Pearson (Biometrika 1934;26[4]:404-413), used underlying event rate of up to 6% in the sugammadex high dose group, based on study results from protocol P06042 (NCT00988065); Test type: Superiority or Other; Difference in incidence = 5.3, 95% CI 2-sided [-0.9 to 10.7] — Difference is Sugammadex 4 mg/kg incidence minus Placebo incidence. Confidence interval calculated using method of Miettinen and Nurminen (Statistics in Medicine 1985;4:213-226)
Statistical Analysis 2: Comparison: Placebo vs Sugammadex 16 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Difference in incidence = 8.1, 95% CI 2-sided [1.7 to 14.2] — Difference is Sugammadex 16 mg/kg incidence minus Placebo incidence. Confidence interval calculated using method of Miettinen and Nurminen(Statistics in Medicine 1985;4:213-226)

2. Secondary Outcome: Percentage of Participants With Adjudicated Anaphylaxis
Description: The investigator or designated clinician performed a THA in each participant at 0.5, 4 and 24 hours after each dose. The THA could also be performed at other times if possible hypersensitivity signs were observed. Each potential hypersensitivity case identified by presence of any sign or symptom in a pre-defined list of hypersensitivity signs and symptoms that were found through the THA was reviewed by an independent, blinded adjudication committee, which determined whether the referred case was a case of anaphylaxis (yes/no) using Sampson Criterion 1 - Acute onset of an illness with involvement of the skin, mucosal tissue or both, and at least one of the following: a) respiratory compromise, b) reduced blood pressure or associated symptoms of end-organ dysfunction (J Allergy Clin Immunol 2006;117:391-397). All AEs occurring in study were reviewed for terms associated with hypersensitivity or anaphylaxis, and could also result in referral to the adjudication committee for evaluation.
Time Frame: Up to approximately 28 days after last dose (approximately 14 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg
Number analyzed (Participants) | 76 | 151 | 148
percentage of participants | 0.0 [0.0 to 4.7] | 0.0 [0.0 to 2.4] | 0.7 [0.0 to 3.7]
Statistical Analysis 1: Comparison: Placebo vs Sugammadex 4 mg/kg; Test type: Superiority or Other; Difference in incidence = 0.0, 95% CI 2-sided [-4.8 to 2.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Sugammadex 16 mg/kg; Test type: Superiority or Other; Difference in incidence = 0.7, 95% CI 2-sided [-4.2 to 3.7] — Difference is Sugammadex 16 mg/kg incidence minus Placebo incidence. Confidence interval calculated using method of Miettinen and Nurminen (Statistics in Medicine 1985;4:213-226)

ADVERSE EVENTS:
Time Frame: Up to approximately 28 days after last dose (approximately 14 weeks)
Description: Analysis performed using APaT population - All randomized participants who received at least one dose of study treatment, with each participant included in arm corresponding to treatment actually received.
Arm/Group | Placebo | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg
Serious Adverse Events (participants affected / at risk) | 2/76 | 2/151 | 1/148
Other Adverse Events (participants affected / at risk) | 18/76 | 50/151 | 75/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Sugammadex 4 mg/kg (N=151) | Sugammadex 16 mg/kg (N=148)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (3)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=76) | Sugammadex 4 mg/kg (N=151) | Sugammadex 16 mg/kg (N=148)
Nausea (Gastrointestinal disorders) | 4 (4) | 16 (21) | 20 (30)
Dysgeusia (Nervous system disorders) | 3 (3) | 11 (15) | 47 (80)
Headache (Nervous system disorders) | 10 (19) | 29 (45) | 30 (52)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 11 (16) | 8 (19)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (11) | 10 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.